CLINICAL TRIAL: NCT03845504
Title: Evaluating the Efficacy and Tolerability of Targeted Transcranial Magnetic Stimulation in Youth
Brief Title: iTBS in Refractory Pediatric Depression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Staffing not available
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 45848
Record Dates: First submitted 2019-02-15; First posted 2019-02-19 (Actual); Results first posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-11

CONDITIONS: Depression
Keywords: depression; transcranial magnetic stimulation; adolescent; treatment refractory
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Open Label (Experimental): Open-label rTMS sessions will occur within ~2 days after the baseline session with daily sessions delivered to left DLPFC over 2-6 weeks.
  Interventions: Device: Intermittent Theta Burst Stimulation

INTERVENTIONS:
Device: Intermittent Theta Burst Stimulation — Stimulation will be administered using the MagVenture MagPro rTMS Research System at currently FDA approved parameters (www.magvitatms.com). The TBS parameters will be 3-pulse 50-Hz bursts given every 200 ms (at 5 Hz) and an intensity of 80% active motor threshold, as measured from the right first dorsal interosseous muscle by a hand-held 700-mm figure-of-eight coil. rTMS will be applied for 9 min delivering a total of 1800 pulses/session.

SUMMARY:
This work will mark the first step in understanding the neural targets for rTMS in youth with difficult to treat depressive symptoms, creating benchmarks for optimizing the safety and efficacy of rTMS for pediatric populations through precision targeting, and encourage funding applications for larger sham- controlled randomized clinical studies.

DETAILED DESCRIPTION:
Problem Statement: Depression is a global health problem with limited novel and targeted solutions. Currently available interventions (medication and psychotherapy) have failed to provide adequate clinical improvement in 40% of adolescents with depression and only produce remission in 30% of youth. There is a clear need to develop better targeted interventions for this growing population of youth.

Specific Aims Aim 1: To examine the efficacy of a targeting strategy to optimize repetitive transcranial magnetic stimulation (rTMS) delivered to the left dorsolateral prefrontal cortex (DLPFC) to reduce depressive symptoms in adolescents between 12-17 years of age. Hypothesis 1: Six weeks of open-label daily intermittent theta-burst stimulation (iTBS) sessions delivered to the left DLPFC will be effective at reducing depressive symptoms between baseline and 10- week follow-up. Hypothesis 2: iTBS over left DLPFC will decrease functional connectivity between left DLPFC and subcallosal cingulate cortex (SCC) and will reduce depression-related hyperconnectivity between nodes of the default mode network (DMN). Hypothesis 3: Higher anti-correlation between left DLPFC and SCC and lower cingulate glutamate concentrations will predict better clinical outcome following iTBS.

Aim 2: To determine the tolerability of iTBS in adolescents between 12-17 years of age. Hypothesis 1: iTBS will be well tolerated without any more than minimal side effects. Hypothesis 2: iTBS will result in sufficient cortical excitability, as measured by 64-channel-EEG pre, during, and post iTBS, to induce an antidepressant effect but not induce seizures or other adverse events.

ELIGIBILITY:
Inclusion Criteria:

* 10 participants ages 12-21 years of age
* with at least moderate to severe depressive symptoms confirmed by the Children's Depression Rating Scale-Revised (CDRS-R>40) or Hamilton Rating Scale for Depression (HRSD-17 ≥ 18)
* able to commit to protocol schedule and provide Informed consent by a legal guardian and assent by a youth participant
* have had at least one prior antidepressant treatment failure with adequate dose and duration

Exclusion Criteria:

* prior neurological diagnosis (neurodevelopmental disorders, strokes/traumatic brain injuries, brain tumor, epilepsy)
* contraindications for TMS or MRI e.g. have any implanted metal
* unstable medical conditions
* acute suicide risk, defined as an attempt in past 6 months that required medical treatment, or history of ≥2 suicide attempts in the past 12 months, or has a clear cut plan for suicide
* pregnancy, suspected pregnancy or not on birth control if sexually active; 6) Inability to locate and quantify a motor threshold
* any factor that the PI determines to be reason for exclusion.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manpreet K Singh, MD MS, Principal Investigator — Associate Professor; Nolan Williams, MD, Principal Investigator — Assistant Professor; Hugh B Solvason, PhD MD, Principal Investigator — Associate Professor
Locations (1):
- Stanford University Pediatric Mood Disorders Program, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
Small pilot study that will be the start of setting up a larger treatment trial that will be publically available. If feasible, results of the pilot study will be published in scientific journals.

REFERENCES:
- [Background] Blumberger DM, Vila-Rodriguez F, Thorpe KE, Feffer K, Noda Y, Giacobbe P, Knyahnytska Y, Kennedy SH, Lam RW, Daskalakis ZJ, Downar J. Effectiveness of theta burst versus high-frequency repetitive transcranial magnetic stimulation in patients with depression (THREE-D): a randomised non-inferiority trial. Lancet. 2018 Apr 28;391(10131):1683-1692. doi: 10.1016/S0140-6736(18)30295-2. Epub 2018 Apr 26. PMID 29726344
- [Background] Oberman LM, Pascual-Leone A, Rotenberg A. Modulation of corticospinal excitability by transcranial magnetic stimulation in children and adolescents with autism spectrum disorder. Front Hum Neurosci. 2014 Aug 13;8:627. doi: 10.3389/fnhum.2014.00627. eCollection 2014. PMID 25165441
- [Background] Wall CA, Croarkin PE, Maroney-Smith MJ, Haugen LM, Baruth JM, Frye MA, Sampson SM, Port JD. Magnetic Resonance Imaging-Guided, Open-Label, High-Frequency Repetitive Transcranial Magnetic Stimulation for Adolescents with Major Depressive Disorder. J Child Adolesc Psychopharmacol. 2016 Sep;26(7):582-9. doi: 10.1089/cap.2015.0217. Epub 2016 Feb 5. PMID 26849202
- [Background] Weigand A, Horn A, Caballero R, Cooke D, Stern AP, Taylor SF, Press D, Pascual-Leone A, Fox MD. Prospective Validation That Subgenual Connectivity Predicts Antidepressant Efficacy of Transcranial Magnetic Stimulation Sites. Biol Psychiatry. 2018 Jul 1;84(1):28-37. doi: 10.1016/j.biopsych.2017.10.028. Epub 2017 Nov 10. PMID 29274805
- [Background] Li CT, Chen MH, Juan CH, Liu RS, Lin WC, Bai YM, Su TP. Effects of prefrontal theta-burst stimulation on brain function in treatment-resistant depression: A randomized sham-controlled neuroimaging study. Brain Stimul. 2018 Sep-Oct;11(5):1054-1062. doi: 10.1016/j.brs.2018.04.014. Epub 2018 Apr 23. PMID 29730251

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4 participants were screened for eligibility, 2 were assigned to the study arm.
Groups:
- Intermittent Theta Burst Stimulation: Daily open-label sessions delivered to left dorsolateral prefrontal cortex (DLPFC) over up to 6 weeks using the MagVenture MagPro repetitive transcranial magnetic stimulation (rTMS) Research System.
Period: Overall Study
Arm/Group | Intermittent Theta Burst Stimulation
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Intermittent Theta Burst Stimulation: Daily open-label sessions delivered to left DLPFC over up to 6 weeks using the MagVenture MagPro rTMS Research System.
Arm/Group | Intermittent Theta Burst Stimulation
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Children's Depression Rating Scale - Revised (CDRS-R) Score From
Description: Standardized assessment to determine depression severity. The CDRS-R total score is the sum of the responses to 17 questions. Each question is graded on a 5- or 7-point scale. Total score ranges from 17-113. In general, higher values of CDRS-R total score represent greater severity of illness. Response to treatment is determined by a ≥ 50% reduction in score from baseline to end of treatment.
Time Frame: Baseline and week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intermittent Theta Burst Stimulation
Number analyzed (Participants) | 2
score on a scale
  Baseline | 73.0 (0.0)
  Change at week 6 | -31.5 (3.5)

2. Secondary Outcome: Change in Hamilton Depression Rating Scale (HDRS-17)
Description: Standardized assessment to determine depression severity. HDRS-17, a clinician-rated measure of depressive symptoms that consists of 17 items rated using a semi-structured interview. Eight of the 17 HDRS-17 items are rated on a 5-point scale (0=absent; 1=doubtful or mild; 2=mild to moderate; 3=moderate to severe; 4=very severe), while the remaining 9 items are rated on a 3-point scale (0=absent; 1=doubtful or mild; 2=clearly present), yielding a minimum total score of 0 (least severe) and a maximum score of 52 (most severe). Response to treatment is determined by a ≥ 50% reduction in score from baseline to end of treatment.
Time Frame: Baseline and week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intermittent Theta Burst Stimulation
Number analyzed (Participants) | 2
score on a scale
  Baseline | 25.5 (0.7)
  Change at week 6 | -11.5 (7.8)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Intermittent Theta Burst Stimulation
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
Early termination led to a small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/04/NCT03845504/Prot_SAP_000.pdf